CLINICAL TRIAL: NCT05736562
Title: Use of Ritual Epre Prenatal Multivitamins to Improve Nutrition Status and Health Outcomes During the Postpartum Period
Brief Title: Use of Ritual Epost Postnatal Multivitamins During the Postpartum Period
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York (Other)
Collaborators: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Xinyin Jiang, Associate professor, City University of New York
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-0670-Brooklyn-2
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Lactation Disorder - Postpartum Condition or Complication; Nutrition, Healthy

STUDY DESIGN:
Intervention Model Description: Women who exclusively breastfeed will be randomized at week 5 postpartum to either receive the Ritual MVI or a blank placebo for 10 weeks.
Who Masked: Participant, Investigator
Masking Description: Neither the participants nor the investigators will know the group assignment. Supplements will be prepared by Ritual and marked with randomly generated ID numbers. Grouping will be revealed by Ritual at end of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ritual Epre (Experimental): This group will receive 2 Ritual Epre multivitamin-mineral supplement pills daily.
  Interventions: Dietary Supplement: Ritual Epre Multimineral-Vitamin Supplement
- Control (Placebo Comparator): This group will receive a blank placebo.
  Interventions: Dietary Supplement: Placebo Control

INTERVENTIONS:
Dietary Supplement: Ritual Epre Multimineral-Vitamin Supplement — The Ritual Epre supplement is a commercially available multivitamin-mineral supplement designed for pregnant and lactating women.
  Arms: Ritual Epre
Dietary Supplement: Placebo Control — This is a customarily designed blank placebo provided by Ritual.
  Arms: Control

SUMMARY:
Multivitamin/multimineral supplements (MVI) provide important nutrition supplement to the diet of pregnant women to cover potential deficiencies and optimize nutrition status of both mom and baby, especially when the diet is suboptimal or nutrient demand is high while absorption is hindered by various factors such as genetic variance and gastrointestinal function. It is, however, largely unknown whether using an MVI during the lactating period helps improve nutrition status of mom and baby. In this double-blind, randomized, controlled trial, the investigators will recruit 7- postpartum women who exclusively breastfeed at week 5 postpartum and randomly assign them to either receive the Ritual MVI which is commercially available or a blank placebo for 10 weeks. A blank placebo is appropriate because there is currently no recommendation or scientific consensus that lactating women who are healthy and eat a normal diet would have improved nutrition status or maternal-infant health outcomes from a nutrition supplement. The investigators will collect blood and breastmilk samples at baseline and end of the study to assess nutrient status. The investigators hypothesize that consumption of a Ritual MVI leads to better nutrition status and biomarkers in maternal-child dyads compared to control.

ELIGIBILITY:
Inclusion Criteria:

* Women are qualified to participate if they are over 10 years of age, having singleton pregnancy, and are exclusively breast feeding and intending to exclusively breast feed for at least 10 more weeks.

Exclusion Criteria:

* Exclusion criteria include diabetes, cardiovascular conditions and liver disease prior to and during pregnancy because these diseases affect metabolism of several nutrients and thus may lead to differences in the MVI intake and nutrient status relationship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Breastmilk folate content | after 10 weeks of intervention
  Breastmilk folate content will be measured
Breastmilk biotin content | after 10 weeks of intervention
  Breastmilk biotin content will be measured.
Postpartum maternal blood folate status | after 10 weeks of intervention
  Blood folate levels will be measured.
Postpartum maternal blood DHA status | after 10 weeks of intervention
  Blood DHA levels will be measured.
Postpartum maternal blood vitamin B12 status | after 10 weeks of intervention
  Blood B12 levels will be measured.
Postpartum maternal blood 3-hydroxyisovaleric acid (3-HIA) status | after 10 weeks of intervention
  3-HIA will be measured
Postpartum stress levels | at week 0 and after 10 weeks of intervention
  The investigators will conduct the Edinburgh Postnatal Depression Scale (EPDS) assessment (maximum score 30, range 0-30, 10 or greater is considered possible depression).
human milk oligosaccharides (HMO) | at week 0 and after 10 weeks of intervention
  HMOs in breastmilk will be measured throughout the study.
Potspartum maternal menaquinone-7 (vitamin K2) status | after 10 weeks of intervention
  undercarboxylated Osteocalcin (ucOC), carboxylated osteocalcin (cOC) and MK-7 will be measured.
Breastmilk MK-7 content | after 10 weeks of intervention
  Breastmilk MK-7 content will be measured.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brooklyn College of City University of New York, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: No